CLINICAL TRIAL: NCT00950157
Title: Testing the Effect of a Caution for Drugs Approved on Surrogate Outcomes Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Attorney General Consumer & Prescriber Education Grant (Other)
Responsible Party: Lisa M. Schwartz, MD, MS, White River Junction VAMC
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 16785
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Risk Communication

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Directive "open question" statement (Experimental): Survey describes the surrogate outcome of the drug along with a directive warning (i.e., stating the issue and why it matters) for drugs shown to improve surrogate outcomes.
  This directive warning mentions that it is not known whether the drug will help patients feel better, and that readers should ask their doctor if there is an available drug shown to improve patient outcomes.
  Interventions: Other: Presentation of information on approval based on a surrogate outcome and levels of caution
- Non-directive open question statement (Experimental): Survey describes the surrogate outcome of the drug along with a non-directive warning (i.e., stating the issue only) for drugs shown to improve surrogate outcomes.
  This non-directive warning mentions only that it is not known whether the drug will help patients feel better.
  Interventions: Other: Presentation of information on approval based on a surrogate outcome and levels of caution
- No open question statement (Experimental): Survey only describes the surrogate outcome of the drug.
  Interventions: Other: Presentation of information on approval based on a surrogate outcome and levels of caution

INTERVENTIONS:
Other: Presentation of information on approval based on a surrogate outcome and levels of caution — Presentation of information that one drug is approved on a surrogate outcome only while another drug has clinical outcomes. Participants are randomized to 1 of 3 caution (e.g. open question") statements: no open question statement, non-directive open question statement or directive open question statement.

SUMMARY:
The purpose of this study is to test whether cautions about the evidence, in this case an "open questions" statement, decreases enthusiasm for drugs that are approved on surrogate outcomes (compared to patient outcomes) alone.

ELIGIBILITY:
Inclusion criteria

* Participants will be randomly selected from a research panel of more than 60,000 U.S. households (Knowledge Networks).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2944 (Actual)
Dates: Start 2009-08; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Hypothetical choice of drug approved on surrogate outcomes vs. drug known to improve patient outcomes | 0 weeks (assessed during intervention)

SECONDARY OUTCOMES:
Strength of opinion (take or refuse doctor's recommendation) for taking the drug approved on surrogate outcomes vs. drug known to improve patient outcomes | 0 weeks (assessed during intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Schwartz, MD, MS, Principal Investigator — White River Junction Veterans Affairs Medical Center; Steven Woloshin, MD, MS, Principal Investigator — White River Junction Veterans Affairs Medical Center

REFERENCES:
- [Derived] Schwartz LM, Woloshin S. Communicating uncertainties about prescription drugs to the public: a national randomized trial. Arch Intern Med. 2011 Sep 12;171(16):1463-8. doi: 10.1001/archinternmed.2011.396. PMID 21911629